CLINICAL TRIAL: NCT01054560
Title: SOLITAIRE™ FR With the Intention For Thrombectomy (SWIFT) Study
Acronym: SWIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWIFT
Record Dates: First submitted 2009-12-10; First posted 2010-01-22 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-08

CONDITIONS: Ischemic Stroke
Keywords: Ischemic Stroke; SOLITAIRE™ Device; SOLITAIRE™; MERCI® Device; MERCI®; Stroke; Ischemic; Mechanical Thrombectomy; Brain; Brain Clot; Brain Artery Revascularization; Recanalization; Brain Stroke; Clot Retriever; Device; Neurosurgery; Neurovascular Intervention; Interventional Neuroradiology; Brain study; neurovascular clinical trial
MeSH Terms: conditions — Ischemic Stroke; Stroke; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOLITAIRE™ Device (Experimental): The SOLITAIRE™ Device (investigational device) is the experimental arm
  Interventions: Device: SOLITAIRE™ Device
- MERCI® Device (Active Comparator): The MERCI® Device (control device) is commercially available.
  Interventions: Device: MERCI® Device

INTERVENTIONS:
Device: SOLITAIRE™ Device — The SOLITAIRE™ Device is the experimental device that will be used in the interventional procedure
  Arms: SOLITAIRE™ Device
Device: MERCI® Device — The MERCI® Device is the control device that will be used in the interventional procedure.
  Arms: MERCI® Device

SUMMARY:
The purpose of this study is to demonstrate substantial equivalence of the SOLITAIRE™ FR Revascularization Device (SOLITAIRE™ Device) with a legally marketed device, MERCI Retrieval System® (MERCI® Device). The study will demonstrate safety and efficacy of the SOLITAIRE™ Device in subjects requiring mechanical thrombectomy diagnosed with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient or patient's legally authorized representative has signed and dated an Informed Consent Form
* Age22-85
* Clinical signs consistent with acute ischemic stroke
* National Institutes of Health Stroke Scale (NIHSS) ≥8and<30
* Thrombolysis in Myocardial Infarction (TIMI) 0 or TIMI 1 flow in the M1 or M2 of middle cerebral artery, internal carotid artery, basilar or vertebral arteries confirmed by angiography that is accessible to the SOLITAIRETM or MERCI® Device
* Patient is able to be treated within 8 hours of stroke symptoms onset with minimum of one deployment of the SOLITAIRETM or MERCI® Device.
* Patient who is ineligible or failed intravenous tissue plasminogen activator (t-PA) therapy given at local institutions or within national practice.
* Patient is willing to conduct follow-up visits

Exclusion Criteria:

* NIHSS > 30 or coma
* Neurological signs that are rapidly improving prior to or at time of treatment
* Females who are pregnant or lactating
* Known serious sensitivity to radiographic contrast agents
* Current participation in another investigation drug or device study
* Uncontrolled hypertension defined as systolic blood pressure > 185 or diastolic blood pressure > 110 that cannot be controlled except with continuous parenteral antihypertensive medication
* Use of warfarin anticoagulation with International Normalized Ratio (INR) > 3.0
* Platelet count < 30,000
* Glucose < 50 mg/dL
* Arterial tortuosity that would prevent the device from reaching the target vessel
* Life expectancy of less than 90 days
* Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of hemorrhage on presentation
* CT showing hypodensity or MR showing hyperintensity involving greater than 1/3 of the middle cerebral artery (MCA) territory (or in other territories, >100 cc of tissue) on presentation
* CT or MRI evidence of mass effect or intracranial tumor (except small meningioma)
* Angiographic evidence of carotid dissection, complete cervical carotid occlusions, or vasculitis

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Saver, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Oregon Stroke Center, Portland, Oregon
  - Multicare Health System, Tacoma, Washington

REFERENCES:
- [Derived] Raychev R, Saver JL, Jahan R, Nogueira RG, Goyal M, Pereira VM, Gralla J, Levy EI, Yavagal DR, Cognard C, Liebeskind DS. The impact of general anesthesia, baseline ASPECTS, time to treatment, and IV tPA on intracranial hemorrhage after neurothrombectomy: pooled analysis of the SWIFT PRIME, SWIFT, and STAR trials. J Neurointerv Surg. 2020 Jan;12(1):2-6. doi: 10.1136/neurintsurg-2019-014898. Epub 2019 Jun 25. PMID 31239326
- [Derived] Coutinho JM, Liebeskind DS, Slater LA, Nogueira RG, Clark W, Davalos A, Bonafe A, Jahan R, Fischer U, Gralla J, Saver JL, Pereira VM. Combined Intravenous Thrombolysis and Thrombectomy vs Thrombectomy Alone for Acute Ischemic Stroke: A Pooled Analysis of the SWIFT and STAR Studies. JAMA Neurol. 2017 Mar 1;74(3):268-274. doi: 10.1001/jamaneurol.2016.5374. PMID 28097310
- [Derived] Kim JT, Jahan R, Saver JL; SWIFT Investigators. Impact of Glucose on Outcomes in Patients Treated With Mechanical Thrombectomy: A Post Hoc Analysis of the Solitaire Flow Restoration With the Intention for Thrombectomy Study. Stroke. 2016 Jan;47(1):120-7. doi: 10.1161/STROKEAHA.115.010753. Epub 2015 Dec 10. PMID 26658447
- [Derived] Sheth SA, Jahan R, Levy EI, Jovin TG, Baxter B, Nogueira RG, Clark W, Budzik R, Zaidat OO, Saver JL; SWIFT Trialists. Rapid learning curve for Solitaire FR stent retriever therapy: evidence from roll-in and randomised patients in the SWIFT trial. J Neurointerv Surg. 2016 Apr;8(4):347-52. doi: 10.1136/neurintsurg-2014-011627. Epub 2015 Feb 12. PMID 25676147
- [Derived] Liebeskind DS, Jahan R, Nogueira RG, Zaidat OO, Saver JL; SWIFT Investigators. Impact of collaterals on successful revascularization in Solitaire FR with the intention for thrombectomy. Stroke. 2014 Jul;45(7):2036-40. doi: 10.1161/STROKEAHA.114.004781. Epub 2014 May 29. PMID 24876081
- [Derived] Liebeskind DS, Jahan R, Nogueira RG, Jovin TG, Lutsep HL, Saver JL; SWIFT Investigators. Serial Alberta Stroke Program early CT score from baseline to 24 hours in Solitaire Flow Restoration with the Intention for Thrombectomy study: a novel surrogate end point for revascularization in acute stroke. Stroke. 2014 Mar;45(3):723-7. doi: 10.1161/STROKEAHA.113.003914. Epub 2014 Feb 13. PMID 24525954
- [Derived] Saver JL, Jahan R, Levy EI, Jovin TG, Baxter B, Nogueira RG, Clark W, Budzik R, Zaidat OO; SWIFT Trialists. Solitaire flow restoration device versus the Merci Retriever in patients with acute ischaemic stroke (SWIFT): a randomised, parallel-group, non-inferiority trial. Lancet. 2012 Oct 6;380(9849):1241-9. doi: 10.1016/S0140-6736(12)61384-1. Epub 2012 Aug 26. PMID 22932715
- See also: American Heart Association - Stroke — http://www.americanheart.org/presenter.jhtml?identifier=3004586
- See also: ev3, Inc. — http://www.ev3.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject enrolled from Feb 2010 to Feb 2011. Subject randomized to Solitaire or Merci by baseline National Institutes of Health Stroke Scale Score.
Pre-assignment Details: Study had Roll-in period. Participating centers in the United States were required to enroll two (2) roll-in subjects prior to the subject randomization. There were a total of 31 roll-in subjects. Only data from the randomized cohort was used for both primary efficacy analysis and the safety endpoint analysis.
Period: Overall Study
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Started | 58 | 55
Completed | 45 | 27
Not Completed | 13 | 28
Not completed — Death | 10 | 21
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOLITAIRE™ Device | MERCI® Device | Total
Number analyzed (Participants) | 58 | 55 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (12.0) | 67.1 (11.1) | 67.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 27 | 57
  Male | 28 | 28 | 56
Region of Enrollment [Number; unit: participants]
  United States | 57 | 54 | 111
  Europe | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Recanalization [Thrombolysis in Myocardial Infarction (TIMI) 2 or 3] Without Symptomatic Intracranial Hemorrhage
Description: Successful arterial recanalization of occluded target vessel measured by Thrombolysis in Myocardial Infarction (TIMI) score of 2 or 3 following the use of the SOLITAIRE™ or MERCI® Device without any symptomatic intracranial hemorrhage and rescue therapy within 3 passes.
  Thrombolysis in Myocardial Infarction (TIMI) score describes the distal flow perfusion and revascularization before and following therapy.
  TIMI 0 - No perfusion (worst outcome) TIMI 1 - Perfusion past the initial occlusion, but no distal branch filling TIMI 2 - Perfusion with incomplete or slow distal branch filling TIMI 3 - Full perfusion with filling of all distal branches (best outcome)
Time Frame: Immediately post treatment
Population: Data was unavailable for two subjects from the randomized Solitaire and one from the randomized Merci cohort. Thus, the Core Lab evaluated data from 56 in the Solitaire FR group and 54 in the Merci group.
Measure: Number; unit: Percent of Subjects
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 56 | 54
Percent of Subjects | 60.7 | 24.1

2. Secondary Outcome: Time to Initial Recanalization
Description: Time from guide catheter placement to first visualization of Thrombolysis in Myocardial Infarction (TIMI) 2 flow
Time Frame: post treatment
Population: Unavailability of data contributed to fewer subjects analyzed compared to the cohort sample size
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 47 | 46
minutes | 47 (37.3) | 58.7 (33.8)

3. Secondary Outcome: Good Neurological Outcome at 30 Days
Description: Good neurological outcome, defined as modified Rankin scale (mRS) ≤ 2, or equal to the prestroke mRS if the prestroke mRS was higher than 2, or National Institutes of Health Stroke Scale (NIHSS) score improvement of 10 points or more
Time Frame: 30 Days Follow-up
Population: Unavailability of data contributed to fewer subjects analyzed compared to the cohort sample size.
Measure: Number; unit: Percent of subjects
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 55 | 51
Percent of subjects | 50.9 | 33.3

4. Secondary Outcome: Good Neurological Outcome 90 Days
Description: as for outcome 3
Time Frame: 90 Days Follow-up
Population: Unavailability of data contributed to fewer subjects analyzed compared to the cohort sample size.
Measure: Number; unit: Percent of subjects
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 55 | 48
Percent of subjects | 58.2 | 33.3

5. Secondary Outcome: Mortality
Description: Rate of Mortality
Time Frame: 90 Days follow-up
Population: Intent-to-treat
Measure: Number; unit: Percentage of subjects
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 58 | 55
Percentage of subjects | 17.2 | 38.2

6. Secondary Outcome: Symptomatic Intracranial Hemorrhage
Description: Symptomatic hemorrhage within 24 hours of procedure. Symptomatic hemorrhages is defined as any parenchymal hematoma 1 (PH1), parenchymal hematoma 2 (PH2), intraparenchymal hemorrhage remote from the ischemic field (RIH), intraventricular hemorrhage (IVH), and subarachnoid hemorrhage (SAH) associated with a worsening of National Institutes of Health Stroke Scale (NIHSS) ≥ 4 within 24hrs.
Time Frame: 24 hours
Population: Intent to treat
Measure: Number; unit: Percentage of subjects
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 58 | 55
Percentage of subjects | 1.7 | 10.9

7. Secondary Outcome: Non-fatal Stroke-related Morbidity
Description: Morbidity data is presented in terms of subjects with permanent deficit as a result of one or more adverse events
Time Frame: 90 Day
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Groups:
- SOLITAIRE™ Device: SOLITAIRE™ Device (investigational device) is the experimental arm
- MERCI® Device: MERCI® Device (control device) is commercially available.
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 58 | 55
percentage of subjects | 43.1 | 32.7

8. Primary Outcome: Study Device-related Serious Adverse Events (SAEs)
Description: Incidence of study device-related Serious Adverse Events (SAEs)
Time Frame: 90 Day
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 58 | 55
percentage of subjects | 9 | 16

9. Primary Outcome: Procedure-related Serious Adverse Events (SAEs)
Description: Incidence of study procedure-related Serious Adverse Events (SAEs)
Time Frame: 90 Day
Population: Intent-to-treat
Measure: Number; unit: percentage of subjects
Arm/Group | SOLITAIRE™ Device | MERCI® Device
Number analyzed (Participants) | 58 | 55
percentage of subjects | 14 | 16

ADVERSE EVENTS:
Time Frame: 90 Days
Description: Independent Clinical Events Committee (CEC) provided independent, unbiased and consistent adjudication for all reportable adverse events.
Groups:
- The SOLITAIRE™ Device: The SOLITAIRE™ Device (investigational device) is the experimental arm
- The MERCI® Device: The MERCI® Device (control device) is commercially available.
Arm/Group | The SOLITAIRE™ Device | The MERCI® Device
Serious Adverse Events (participants affected / at risk) | 49/58 | 44/55
Other Adverse Events (participants affected / at risk) | 37/58 | 30/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The SOLITAIRE™ Device (N=58) | The MERCI® Device (N=55)
Anaemia (Blood and lymphatic system disorders) | 9 (10) | 4 (4)
Atrial Fibrillation (Cardiac disorders) | 11 (12) | 4 (4)
Retinal Artery Occlusion (Eye disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 2 (2) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 2 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Air embolism (Vascular disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1) | 0 (0)
Artrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardyia (Cardiac disorders) | 1 (1) | 2 (2)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 3 (4)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Device breakage (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 6 (6)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) | 5 (5)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Clostridal infection (Infections and infestations) | 1 (1) | 1 (1)
Bacterial disease carrier (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Procedural hypertension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral nerve injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 1 (1) | 1 (1)
Echocardiogram abnormal (Investigations) | 2 (2) | 0 (0)
Lipids increased (Investigations) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0)
Blood creatinine (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral gas embolism (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral haematoma (Nervous system disorders) | 5 (5) | 8 (8)
Cerebrovascular accident (Nervous system disorders) | 7 (7) | 13 (13)
Cerebrovascular spasm (Nervous system disorders) | 3 (3) | 4 (4)
Convulsion (Nervous system disorders) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic cerebral infarction (Nervous system disorders) | 4 (4) | 3 (3)
Intracranial pressure increased (Nervous system disorders) | 2 (2) | 2 (2)
Intraventricular haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 7 (7)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 3 (3) | 7 (7)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (8)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 2 (2)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 6 (7) | 5 (5)
Intra-abdominal haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Vasospasm (Vascular disorders) | 3 (3) | 3 (3)
Vessel perforation (Vascular disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Catheter Site Haemorrhage (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | The SOLITAIRE™ Device (N=58) | The MERCI® Device (N=55)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Eye oedema (Eye disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 3 (3)
Unintentional medical device removal by patient (General disorders) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Clostridial infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 12 (12) | 6 (7)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Differential white blood cell count abnormal (Investigations) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (5)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper extremity mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery dissection (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhagic cerebral infarction (Nervous system disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 6 (6) | 2 (2)
Intracranial pressure increased (Nervous system disorders) | 2 (2) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Muscle spasticity (Nervous system disorders) | 1 (1) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hpoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 2 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Labile blood pressure (Vascular disorders) | 1 (1) | 0 (0)
Thromophlebitis superficial (Vascular disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Physician shall not make any publication without providing Sponsor 30 days notice.If Sponsor determines that the proposed publication contains confidential information, Sponsor may require the delay of publication for a period of time not to exceed 90 days and may require that any confidential information be removed from the publication. Sponsor may also require Physician to delay publication until any factual errors or inaccuracies in the publication are corrected.